CLINICAL TRIAL: NCT01314651
Title: Efficacy of Behavioral Insomnia Treatment for Chronic Migraine: A Randomized Controlled Pilot Study
Brief Title: Efficacy of Behavioral Insomnia Treatment for Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Riche (Other)
Collaborators: Migraine Research Foundation (Other); The Oxford Neurology Clinic (Unknown)
Responsible Party: Sponsor-Investigator, Daniel Riche, University of Mississippi Clinical Trials and FDA Administrator, University of Mississippi, Oxford
Organization: University of Mississippi, Oxford (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMO-0002
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Migraine; Insomnia
Keywords: Migraine Disorders; Chronic migraine; Insomnia; Behavioral sleep management
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Management (Experimental): Instructions in stimulus control and sleep restriction.
  Interventions: Behavioral: Stimulus Control and Sleep Restriction
- Lifestyle Modification (Sham Comparator): Instructions to change general lifestyle habits (maintain consistent liquid consumption, range of motion exercises, etc.)
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Behavioral: Stimulus Control and Sleep Restriction — 5 instructions in stimulus control and individually-tailored sleep restriction
  Arms: Sleep Management
Behavioral: Lifestyle Modification — 5 instructions in changing general lifestyle habits (maintaining consistent liquid intake, range of motion exercises, eating a serving of protein in the morning, etc.)
  Arms: Lifestyle Modification

SUMMARY:
The purpose of this study is to test the efficacy of a brief behavioral insomnia intervention in reducing headache frequency and severity among patients with chronic migraine and insomnia. It is hypothesized that this intervention will produce greater changes in headache frequency and severity than will a comparison treatment involving non-sleep-specific general lifestyle modifications.

DETAILED DESCRIPTION:
Chronic migraine (occurring 15 or more days per month) is a disabling disorder that engenders significant personal suffering and healthcare costs. Frequently, individuals with chronic migraine also suffer from symptoms of insomnia, the regulation of which has been shown to improve migraine. A variety of effective and well-validated behavioral treatments exist to reduce symptoms of insomnia but have not been widely applied to migraine patients. The goal of this study is to pilot test and compare the efficacy of 2 different behavioral (non-medication) treatments for chronic migraine, one of which addresses insomnia symptoms and one of which addresses general lifestyle changes, on headache and sleep parameters. Patients will be adults (18-65) diagnosed with chronic migraine and insomnia at the Oxford Neurology Clinic when they present for routine medical appointments. They will be maintained on usual medical care and referred to the Psychological Services Center for collection of baseline data and administration of the behavioral interventions. At baseline participants will be administered a structured interview and questionnaires pertaining to headache symptoms, sleep problems, and depression/anxiety. They will keep a daily diary of headache variables for 2 weeks and wear an actigraph on their wrist during baseline. Patients will be randomly assigned to receive either the a treatment focused on modifying general lifestyle behaviors (Lifestyle Modification; a replication of the instructions from Calhoun and Ford, 2007) or making changes to their sleep behaviors (Sleep Management) for 3 brief (20-30 min) sessions, spaced 2 weeks apart. Treatments will entail education/rationale about the intervention and a review of a set of instructions unique to each condition. Subsequent sessions will ensure compliance with the respective instructions. Daily monitoring of headache symptoms will continue throughout the trial. Participants will complete the aforementioned questionnaires at 2 posttreatment follow-up visits and wear the actigraph again for 2 week periods surrounding the 2 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 diagnosed with chronic migraine (15 or more days with headache per month, most of which must be migraine) and insomnia who present for routine medical care for migraine.

Exclusion Criteria:

* Currently pregnant or breastfeeding, being unable to read or speak English at a 6th grade level, alcohol or substance abuse or dependence, bipolar disorder or seizure disorder, psychiatric hospitalization within the last year, medication overuse headache, and patients not stable on current migraine medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Headache frequency | 2 weeks post-treatment, 6 weeks post-treatment

SECONDARY OUTCOMES:
Headache severity | 2 weeks post-treatment, 6 weeks post-treatment
Headache-related disability | 2 weeks post-treatment; 6 weeks post-treatment
Total Sleep Time | 2 weeks post-treatment; 6 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Smitherman, Ph.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Psychological Services Center, University, Mississippi, United States

REFERENCES:
- [Derived] Smitherman TA, Walters AB, Davis RE, Ambrose CE, Roland M, Houle TT, Rains JC. Randomized Controlled Pilot Trial of Behavioral Insomnia Treatment for Chronic Migraine With Comorbid Insomnia. Headache. 2016 Feb;56(2):276-91. doi: 10.1111/head.12760. Epub 2016 Jan 27. PMID 26813845